CLINICAL TRIAL: NCT05501444
Title: Antiperspirant in the Treatment of Residual Limp Hyperhidrosis for Prosthetic Users: a Pilot Study
Brief Title: Antiperspirant in the Treatment of Residual Limp Hyperhidrosis for Prosthetic Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sophies Minde Ortopedi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FoU_2022_Hyperhidrosis
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Hyperhidrosis; Residual Limbs
Keywords: Lower limb amputation; Hyperhidrosis; Prosthetic users; Aluminum chloride; Sweating
MeSH Terms: conditions — Hyperhidrosis | interventions — Antiperspirants

STUDY DESIGN:
Intervention Model Description: The project is carried out as a pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effect of antiperspirant (Experimental): Aluminium chloride 15 percent
  Interventions: Other: Topical antiperspirant

INTERVENTIONS:
Other: Topical antiperspirant — The participants will be instructed to use topical antiperspirant (aluminum chloride, 15 percent every evening for four weeks. The PI will contact the participants every week. If the participant experiences that antiperspirant have an effect, the use of antiperspirant will be reduced from daily use to 3 times a week.

SUMMARY:
The aim of the present pilot study is to evaluate the effect of antiperspirant to treat residual limb hyperhidrosis with the emphasis on the utility of the iodine-starch test to identify the location of the sweating.

DETAILED DESCRIPTION:
Many persons with lower limb amputation report that they have major problems with sweating (hyperhidrosis) on the stump in connection with prosthetic use. Despite the frequency and the negative effect of sweating for prosthetic users, there is a lack of evidence on how the sweating should be examined and treated. In the dermatological literature, the guidelines recommend the use of topical antiperspirants such as aluminum chloride as first-line treatment. No studies have previously been published evaluating the effect of antiperspirant on prosthetic users.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years,
2. used a prosthetic for at least 1 year,
3. HDSS score of ≥ 2,
4. use the prosthetic daily and be able to walk for a minimum of 10 minutes.

Exclusion Criteria:

1. Open wounds on the stump,
2. Known sensitivity or allergy to iodine and/or starch,
3. Known sensitivity to antiperspirant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Hyperhidrosis Disease Severity Scale (HDSS) | Four weeks
  The HDSS is a short single-item scale that is scored from 1-4 and provides a qualitative measure of the severity of sweating based on the extent to which sweating affects daily activities.
Sweating Intensity Visual Scale (SIVS) | Four weeks
  In connection with the Minor test, it is also recommended to use the Sweating Intensity Visual Scale (SIVS) in order to provide a more objective and standardized interpretation of the results of the Minor test. SIVS is graded on a scale from 0-V (Grade 0= minimal or no sweating, Grade I = initial, discrete sweating, Grade II = mild sweating, Grade III = moderate sweating, Grade IV = intense sweating, and Grade V= oversweating)

SECONDARY OUTCOMES:
Numerical Ranking Scale (NRS 100) | Four weeks
  Numerical Ranking Scale (NRS 100) (with 0 as low and 100 as high) is used to investigate the following question:
  * How much sweating do you experience on the stump?
  * How much does sweating affect your function?
  * How much does sweating reduce your quality of life?
  * How much does sweating affect walking related to instability?
  * How much does sweating affect your activity level?
  * How much does sweating affect your skin quality on the stump

CONTACTS AND LOCATIONS:
Overall Officials: Jette Schack, PhD, Principal Investigator — Sophies Minde Ortopedi
Locations (1):
- Sophies Minde Ortopdi AS, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No